CLINICAL TRIAL: NCT06927284
Title: Effects of Neurocognitive Therapy With and Without Soft Robotic Hand on Hand Function in Sub-acute Stroke
Brief Title: Effects Of Neurocognitive Therapy With And Without Soft Robotic Hand On Hand Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0217 Shazia
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Hand Function; Cognition
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and outcome assessors will be kept blinded about the intervention which the patients will be going to recieve.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurocognitive Therapy with Soft Robotic Hand based (Experimental): Neurocognitive therapy group with soft robotic hand for 30 minutes along routine physical therapy for 15 minutes , the participants will be blindfolded during the exercises and ask to concentrate on sensing the position of the limb and hand Opening and closing of the soft robotic glove is controlled by the hand control switch .Treatment session of 45 minutes will be given 3 times a week for 12 week.
  Interventions: Other: Neurocognitive Therapy without Soft Robotic Hand
- Neurocognitive Therapy without Soft Robotic Hand based (Experimental): Neurocognitive therapy group without soft robotic hand for 30 minutes along routine physical therapy for 15 minutes , the participants will be blindfolded during the exercises and ask to concentrate on sensing the position of the limb and hand Opening and closing of the soft robotic glove is controlled by the hand control switch .Treatment session of 45 minutes will be given 3 times a week for 12 week.
  Interventions: Other: Neurocognitive Therapy with Soft Robotic Hand

INTERVENTIONS:
Other: Neurocognitive Therapy with Soft Robotic Hand — There will be 23 participants received Neurocognitive Therapy with soft robotic hand . Total 45 minutes session will be provided to patient including 15 minutes of routine physical therapy training for upper limb. The following hand exercises will be performed . Passive localization, passive identification, and active object exploration .For localization placed a part of the patient's limb, typically the fingertip, on one external object (e.g. sand paper, toothpick, sponge, paint brush, cotton ball, pencil, eraser ) and for identification water bottle, sponge, toothpaste tube, electrical plug, plastic ball, paper cup, tape roll, metal bolt with nut, tape roll . During active exploration the The training object repositioned, and another object of a different shape or size offered (water bottle, water bottle with ice in it, sponge. The blindfolded patient then used his effected hand to explore different objects and asked to identify each object with soft robotic hand.
  Arms: Neurocognitive Therapy without Soft Robotic Hand based
Other: Neurocognitive Therapy without Soft Robotic Hand — There will be 23 participants received Neurocognitive Therapy without soft robotic hand . Total 45 minutes session will be provided to patient including 15 minutes of routine physical therapy training for upper limb. The following hand exercises will be performed . Passive localization, passive identification, and active object exploration .For localization placed a part of the patient's limb, typically the fingertip, on one external object (e.g. sand paper, toothpick, sponge, paint brush, cotton ball, pencil, eraser ) and for identification water bottle, sponge, toothpaste tube, electrical plug, plastic ball, paper cup, tape roll, metal bolt with nut, tape roll . During active exploration the The training object will be repositioned, and another object of a different shape or size will be offered (water bottle, water bottle with ice in it, sponge. The blindfolded patient then used his effected hand to explore different objects and asked to identify each object .
  Arms: Neurocognitive Therapy with Soft Robotic Hand based

SUMMARY:
To determine the effect of neurocognitive therapy with and without a soft robotic hand on manual ability, dexterity, strength, spasticity and upper limb function in sub-acute stroke.

DETAILED DESCRIPTION:
Stroke is a global disease with high death rate and high disability caused by motor cortical damage. According to the calculations, there were approximately 13.68 million new increased stroke patients all over the world a year and about 70% of survivors had diﬀerent degrees of upper limb and hand movement dysfunction .The recovery rate of patients' motor function mainly depends on rehabilitation training. Therefore, due to individual diﬀerence of patients. Neurocognitive therapy is an effective therapy to improve and increase cognitive, sensory and motor function of upper limb. Robotic hand also help the function of weak hand muscle. Neurocognitive therapy with a robotic hand will have the potential to offer targeted, precise, and adaptable interventions, possibly increase the rehabilitation process compared to both interventions alone. Evaluating their relative efficacy will aid in refining and tailoring rehabilitation strategies for individuals recovering from acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* Participants of Post stroke patients (6-12 weeks )
* Participants with Spasticity < 2 on modified Ashworth scale.
* Participants with first ever stroke.
* Participants with normal cognition > 24 on MoCA
* Participants must be able to provide informed consent
* Hemiparesis with arm motor deficit as assessed by with NIHSS >1(14)

Exclusion Criteria:

* Participants who have a history of significant neurological or orthopedic disorders, other than stroke, that could interfere with upper limb motor or sensory recovery.
* Participants who have altered state of consciousness, severe aphasia, severe cognitive deficit.
* Participants who have severe pathologies of traumatic and or rheumatic nature, severe pain in effected arm (>5 on visual analog scale for pain) .
* Participants who have active pacemakers and other active implants.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Montreal cognitive assessment (MoCA): (cognition) | 12 Weeks
  The Montreal Cognitive Assessment (MoCA) is a one-page, 30-point cognitive screening measurement scale that takes about 10 minutes to administer. There are 12 subtasks in the MoCA test that include memory, visuospatial orientation, executive functioning, phonemic fluency, and two-item abstract thinking task, attention, concentration, and working memory, language, orientation to time and place. A score of 26 is a cutoff score to differentiate between normal and abnormal. Inter-rater Reliability (0.96) Cronbach's alpha .Change will be measured from baseline to 12 weeks.
Barthel Index (basic activities of daily living) | 12 Weeks
  The BI is a measure of functional status whose validity when used on a general population of older people has been shown . The BI uses 10 items . Of the 10 items, two (bathing and grooming) are rated on a two-point scale of 0 and 1, six (feeding, dressing, bowels, bladder, toilet use and stairs) on a three-point scale of 0, 1 and 2 and the last two items (transfers and mobility) are rated on a four-point scale of 0, 1, 2 and 3. Change will be measured from baseline to 12 weeks.
Modified Ashworth Scale (MAS)( spasticity level of the upper limb) | 12 Weeks
  The original Ashworth scale was a 5 point numerical scale that graded spasticity from 0 to 4, with 0 being no resistance and 4 being a limb rigid in flexion or extension. In 1987, while performing a study to exam interrater reliability of manual tests of elbow flexor muscle spasticity, Bohannon and Smith modified the Ashworth scale by adding 1+ to the scale to increase sensitivity. Change will be measured from baseline to 12 weeks.
Erasmus MC Nottingham Sensory Assessment (ErNSA) (sensation and proprioceptive) | 12 Weeks
  The ErNSA is a specialized assessment tool designed to evaluate tactile sensation and proprioceptive ability in the upper limb. It consists of various subtests that provide a detailed examination of sensory function, contributing valuable insights into the sensory recovery post stroke of the upper limb).Change will be measured from bassline to 12 weeks.
) Action Research Arm Test (grasping, grip- ping, pinching) | 12 Weeks
  The ARAT is a hierarchical scale for the evaluation of arm-hand capacity. It consists of 19 functional items that are divided into 4 subtests: grasp, pinch, grip, and gross motor function. A total score of 57 indicates normative performance. The reliability and validity of the ARAT for patients with stroke have been established. on ARAT scores and subsequently classified into 5 different categories: 0 to 10 points as no capacity, 11 to 21 points as poor capacity, 22 to 42 points as limited capacity, 43 to 54 points as notable capacity, and 55 to 57 points as full capacity. Change will be measured from baseline to 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD*, Principal Investigator — Riphah International University; Shazia Abdul Mateen, Study Chair — Riphah International University
Locations (1):
- Sheikh Zayad Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No